CLINICAL TRIAL: NCT06338501
Title: Assessment of Heart Rate Variability, Performance and Dehydration in Muay Thai Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77325224.4.0000.5235
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Nervous System Diseases; Dehydration
MeSH Terms: conditions — Nervous System Diseases; Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Exercise (Experimental): 30 functional specific exercises for muaythai athletes. Nutrition Control HRV quantify.
  Interventions: Other: Specifical Functional Training Exercises

INTERVENTIONS:
Other: Specifical Functional Training Exercises — Strength Training: Include compound exercises like squats, deadlifts, lunges, and bench presses to build overall strength and muscle mass. Focus on functional movements that mimic the actions used in Muay Thai.
  Core Stability Exercises: A strong core is essential for generating power and maintaining balance during strikes and defensive maneuvers.
  Plyometric Training: Jumping exercises such as box jumps, squat jumps, and split jumps help improve explosive power and enhance muscular endurance, crucial for delivering swift and powerful strikes.
  Flexibility and Mobility Training: Incorporate stretching exercises to improve flexibility, joint range of motion, and prevent injuries.
  Interval Training: Perform high-intensity interval training (HIIT) sessions that combine cardiovascular exercises.

SUMMARY:
Known as "Thai boxing," Muay Thai utilizes a combination of upper limb strikes (such as punches and elbow strikes) as well as lower limb strikes (such as kicks and knee strikes), and is thus referred to as the "art of eight limbs." It is practiced worldwide and is a prominent discipline in many mixed martial arts (MMA) training camps. In this sport, training load control involves monitoring and adjusting the quantity and intensity of training according to each athlete's capacity. In the context of combat sports, such as Muay Thai, heart rate variability (HRV) and assessment of body composition by bioelectrical impedance analysis can be used as tools to evaluate training responses. Additionally, HRV can also serve as a tool for assessing recovery after training or competition. If HRV does not return to baseline after training or competition, it may be a sign that the athlete is not fully recovered and may need more time to recuperate before returning to training or competition. Due to the absence of studies in the literature that have assessed a possible association between HRV and dehydration and rehydration processes in amateur Muay Thai athletes, it becomes essential to evaluate this correlation. Given the growing interest in practicing Muay Thai in gyms, assessing the sympathetic-vagal balance, body composition, and performance of these athletes becomes of utmost importance. Therefore, the aim of this study is to investigate the relationship between dehydration indicators, HRV parameters, and performance in the frequency speed kick test (FSKT). Participants will be assessed before and after an eight-week training program, conducted three times a week. Assessments will include resting HRV measurement and FSKT; in addition, bioimpedance will be used to estimate the body composition of participants pre- and post-training. It is expected that the results will reveal changes in HRV, performance, and body composition of the athletes after training.

ELIGIBILITY:
Inclusion Criteria:

- 1. Amateur Muay Thai athletes from the city of Curitiba and metropolitan region, aged ≥ 18 years old, male.

2. Amateur Muay Thai athletes for a minimum period of 6 months.

Exclusion Criteria:

* 1. Pregnant women. 2. Uncontrolled high blood pressure. 3. Inability to perform performance tests 4. Interrupting any test spontaneously

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
HRV during specifical physical test | 1 year
  Measurement of HRV obtained during the FSKT protocol, pre and post-training of 8 weeks specific conditioning and strength for Muay Thai and nutritional intervention.

SECONDARY OUTCOMES:
Correlation with BIA analysis, HRV and Specific Physical Test | 1 year
  Based on the results obtained through the Bioelectrical Impedance Analysis (BIA) test, the existence of potentially significant correlations between these measurements and the activity of the autonomic nervous system, specifically sympathetic-vagal regulation, is being investigated, assessed through analysis of Heart Rate Variability (HRV).

IPD SHARING:
Plan to Share IPD: No